CLINICAL TRIAL: NCT06266169
Title: Application of Spectral Methods to Assess the Potential of Gametes and Embryos, as Well as Human Reproductive Capabilities
Brief Title: Application of Spectral Methods to Assess Gametes, Embryos, and Human Reproductive Capabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Family Planning Center of Women's Welfare Clinic #44 of Pushkin District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: fpc-2023-ivf-01
Record Dates: First submitted 2024-02-01; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: For the retrospective (observational) stage of the study:
  Embryos: 424 samples of the culture medium used from individually cultured blastocysts that were fresh and frozen before transferring a single embryo from the institution's internal biobank. Each sample is attributed based on the presence or absence of progressing pregnancy after transfer at 12-14 weeks.
  Semen: 340 samples of sperm from the internal biobank of couples undergoing ICSI, each sample is attributed based on the success or failure of the embryological stage.
  Endometrium: 300 samples of luminescent and visible spectra of patients' endometrium undergoing embryo transfer, each sample is attributed based on the presence or absence of ongoing pregnancy after transfer.
  For the prospective (interventional) stage of the study:
  For each object of study, the size of the dataset for prospective testing can only be determined after passing the observational part of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): People undergoing IVF treatment with developed medical decisions support models
  Interventions: Other: making artificial intelligence based decisions of gamete, embryo and endometrial potential
- control (No Intervention): People undergoing IVF treatment without developed medical decisions support models

INTERVENTIONS:
Other: making artificial intelligence based decisions of gamete, embryo and endometrial potential — The method of Raman spectroscopy is based on the registration of inelastic scattering of photons. Each compound has its own spectral pattern when using a certain type of monochromatic radiation (laser). With this method, it is possible to obtain metabolic fingerprints from the objects being studied. Luminescent spectroscopy is a type of spectroscopy used to register emission from objects that occurred after absorbing the exciting (primary) radiation. Spectrophotometry is the detection of radiation in the visible area of the spectrum. Raman spectroscopy is used for the spent medium and semen to build artificial intelligence model and make prognosis of function for each object. For endometrium, luminescent spectroscopy and spectrophotometry are used to build the model and test its clinical relevance
  Arms: intervention

SUMMARY:
Relevance of the research topic: At present, in the world, a kind of "plateau" in the efficiency of assisted reproductive technologies has been achieved, which ensures a birth rate of 30% per embryo transfer. At the same time, a relatively high (15-20%) and stable rate of miscarriages is preserved. Until now, no effective methods for assessing the potential of gametes and embryos, as well as human reproductive capabilities, have been offered. In these conditions, to increase the rate of births after IVF, clinicians have to increase the number of transferred embryos at a time, however, this leads to a sharp increase in complications of IVF, such as multiple pregnancy. In addition, until today, the clinical effectiveness of assessing the potential of endometrium using gene expression determination methods has not been shown. Therefore, to ensure the effectiveness and safety of infertility treatment, it is necessary to develop methods for predicting the potential of gametes and embryos, as well as human reproductive capabilities. For this purpose, the investigators assume to use Raman spectroscopy of the environment obtained from the objects of research, as well as fluorescent spectroscopy of endometrium. The objects of the research are gametes (spermatozoa) and embryos, used culture medium, endometrium. The subject of the study is the set of factors, that exists in the objects of research and their ability to determine the outcomes of infertility treatment.

DETAILED DESCRIPTION:
The goal of the planned work is to build a system for assessing and predicting the potential of gametes and embryos, as well as human reproductive capabilities, based on spectral data obtained from the objects of investigation, followed by prospective validation of the developed system. The study protocol consists of a retrospective and prospective stages. The task of the retrospective stage is to study gametes, embryos, and endometrium using the declared methods and build a machine learning model, determine the predictive capabilities of the obtained models. The task of the prospective stage is to determine the practical efficiency of applying models for making clinically significant decisions in infertility treatment with IVF. Hypothesis of the study: at the moment, a large number of approaches and protocols for deselecting and selecting embryos / gametes, assessing endometrial receptivity has been proposed. Approaches related to deselection are mainly based on determining the genetic constitution (aneuploidy) of the investigated object. However, there are no models linking such testing results and the outcome of infertility treatment with clinically significant effectiveness. There are many publications when, after transferring aneuploid embryos, pregnancy develops with a healthy fetus. It is known that the concordance of aneuploidy test results between the internal cell mass and trophoblasts is about 60%. Moreover, when using PGT-a, the birth rate among women with a single available blastocyst is reduced twice. Approaches related to selection, i.e. predicting a positive outcome of treatment, are built on morphological, morphometric, metabolic, and gene expression approaches. However, their effectiveness either has not been proven, or has (if it has) relatively low predictive importance. This is due to the fact that, from the point of modern views on reproductive biology, for the occurrence and development of successful pregnancy, it is necessary to combine factors that belong to gametes, embryos, and the maternal organism. Also, other undetectable technical or other circumstances may play a role in influencing the chance of ongoing pregnancy. Therefore, for effective prediction of a positive outcome, it is necessary to develop and apply complex models that take into account variables from different sources, from all parties involved. However, there will always be additional variability, caused by a series of unspecified or difficult to specify factors, which makes the task of such prediction quite challenging. In this connection, predicting a negative outcome of treatment (deselecting objects) seems more sensible, as it is entirely feasible for cases, where the cause of the negative outcome is attributable to this object (for example, the state of the embryo). This will not only optimize patient care protocols (for example, not to transfer obviously incapable to implant embryos), but also determine the possible cause of the negative outcome in each specific case, and in a population scale determine the share of variability of the phenomenon (development of ongoing pregnancy), which may be related to a specific object. The last one is necessary for adequate development and testing of new therapeutic and diagnostic methods

ELIGIBILITY:
Inclusion Criteria:

* Embryos: embryos that have reached the blastocyst stage
* Sperm: samples used for IVF during infertility treatment
* Endometrium: endometrial spectra in cases where an embryo transfer was performed into the uterus

Exclusion Criteria:

* For all groups: ectopic pregnancy
* Embryos: presence of only one blastocyst, and that embryo prognosed by the model as negative
* Sperm: a cycle where less than 3 oocytes suitable for fertilization were obtained; total pathological fertilization; 60% or more immature oocytes at the time of fertilization registration

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1064 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Embryonic model performance | 14 weeks
  Positive predictive value for negative outcomes of single embryo transfers (%)
Gamete model performance | 2 weeks
  Positive predictive value for cycles with impaired embryo development in vitro (%)
Endometrial model performance | 14 weeks
  Positive predictive value for negative outcomes of single embryo transfers (%)
Embryonic model clinical efficiency | 14 weeks
  Ongoing pregnancy rate per single embryo transfer (%)
Endometrial model clinical efficiency | 14 weeks
  Ongoing pregnancy rate per single embryo transfer (%)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Gryaznov, Principal Investigator — Family planning center of SPB SBHI "Maternity welfare clinic" #44 of Pushkin district
Locations (1):
- Family planning center, Saint Petersburg, Pushkin, Russia

IPD SHARING:
Plan to Share IPD: No